CLINICAL TRIAL: NCT01301287
Title: The Effect of Chlorella on Glycemic Control of Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardinal Tien Hospital (Other)
Collaborators: Tri-Service General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTH-96-2-028
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (1):
- Chlorella (Experimental)
  Interventions: Drug: Chlorella

INTERVENTIONS:
Drug: Chlorella

SUMMARY:
Chlorella, a type of unicellular fresh water algae, has been a popular foodstuff in Asia, especially in Taiwan. Recent studies have shown the hypoglycemic effects of Chlorella through increasing glucose uptake in the liver and muscle, lowering serum free fatty acid levels, or activation of PPAR gamma receptor. However, the hypoglycemic effect in diabetic patients have not been studied. In order to clarify the hypoglycemic effects and mechanism of Chlorella in diabetic patients, the investigators conducted a 12-week randomized, double-blind, placebo-control trial on diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* type 2 diabetes with less than 2 kinds of oral antidiabetes drugs
* Hba1c: 7.0-9.0

Exclusion Criteria:

* type 1 diabetes
* pregnancy
* acute infectious disease
* autoimmune disease
* hemodynamic unstable

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01

PRIMARY OUTCOMES:
HbA1c | 12 weeks

SECONDARY OUTCOMES:
Insulin concentration during oral glucose tolerance test | 12 weeks
  All subjects received the first oral glucose tolerance test before intervention(week 0), and the second oral glucose tolerance test on week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Dee Pei, MD, Principal Investigator — Cardinal Tien Hospital 362, Chung Cheng Rd., Hsintien Taipei County 23137 Taiwan R.O.C.
Locations (1):
- Cardinal Tien Hospital, New Taipei City, Taiwan